CLINICAL TRIAL: NCT05521516
Title: Percutaneous Auricular Neuromodulation for Postoperative Analgesia: A Randomized, Participant- and Observer-Masked, Sham-Controlled Pilot Study
Brief Title: Percutaneous Auricular Neuromodulation for Postoperative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Auricular NeuromodulationPilot
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Parallel Assignment: Randomized, Triple-Masked, Placebo-Controlled, Parallel-Arm Human Subjects Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Investigational Drug Service will create the randomization tables and provide the investigators with the appropriate device (active or sham), leaving all participants, investigators, and the statistician masked to treatment group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active Percutaneous Auricular Neuromodulation with NSS-2 Bridge (Active Comparator): Application of 5 days of percutaneous auricular Neuromodulation with NSS-2 Bridge device
  Interventions: Device: Active Percutaneous Auricular Neuromodulation with NSS-2 Bridge
- Sham Treatment (Sham Comparator): Application of 5 days of a nonfunctional sham device
  Interventions: Device: Sham Treatment

INTERVENTIONS:
Device: Active Percutaneous Auricular Neuromodulation with NSS-2 Bridge — Application of 5 days of percutaneous auricular neuromodulation with NSS-2 Bridge device
  Arms: Active Percutaneous Auricular Neuromodulation with NSS-2 Bridge
Device: Sham Treatment — Application of 5 days of a nonfunctional sham device
  Other Names: Placebo
  Arms: Sham Treatment

SUMMARY:
The moderate-to-severe pain many patients experience following surgery is often treated with opioids, which are associated with side effects such as nausea/vomiting, sedation, and respiratory depression (and a risk of abuse, dependence, and diversion). Potent site-specific analgesia with fewer side effects may be provided with peripheral nerve blocks. However, these too have limitations such as a duration of action measured in hours, while the pain from surgery is usually measured in days or weeks. Peripheral nerve stimulation or "neuromodulation" is an alternative method of pain control involving the introduction of electrical current to stimulate various nerves that do not carry pain sensations, but which then decreases communication between pain fibers and the spinal cord and/or brain. Placing small electrodes specifically in the area of the ear is called "auricular neuromodulation" and is theorized to function by stimulating various cranial and peripheral nerves that influence a part of the brain called the "limbic system" which is involved with many aspects of behavior including responses to stress. A device that delivers auricular neuromodulation, the "Bridge" system, is approved by the United States Food and Drug Administration for use to reduce symptoms associated with opioid withdrawal for up to 5 days. However, one prospective and two published retrospective studies suggest that it may provide postoperative analgesia as well. The device itself is relatively simple to apply; has few contraindications, side effects, or adverse events; and has no potential for dependence, abuse, or diversion. Therefore, it has the potential to concurrently improve analgesia and decrease or even negate opioid requirements following surgery, only without the limitations of opioids and peripheral nerve blocks. The purpose of this pilot study is to explore the possibility of treating postoperative pain with percutaneous auricular neuromodulation, optimize the study protocol, and estimate the treatment effect in preparation for developing a subsequent definitive clinical trial.

DETAILED DESCRIPTION:
The proposed study will be a randomized, participant- and observer-masked, sham-controlled, parallel-arm, human participants pilot study with two primary aims:

Specific Aim 1: To determine the feasibility and optimize the protocol for a subsequent clinical trial that will compare the addition of percutaneous auricular neuromodulation to usual and customary analgesia following moderate-to-severely painful surgical procedures.

Specific Aim 2: To estimate the treatment effect of adding percutaneous auricular neuromodulation to usual and customary analgesia on pain and opioid consumption following various surgical procedures. This will provide an idea of the optimal surgical procedures amenable to this analgesic technique and allow determination of the required sample size of a subsequent definitive clinical trial.

Hypothesis 1: Auricular neuromodulation decreases pain in the 5 days following moderate-to-severely painful surgical procedures currently treated with a single-injection peripheral nerve block.

Hypothesis 2: Auricular neuromodulation decreases opioid use in the 5 days following moderate-to-severely painful surgical procedures currently treated with a single-injection peripheral nerve block.

This will be a single-center (UCSD), randomized, participant- and observer-masked, sham-controlled, parallel-arm human participants pilot study.

Enrollment. Participants will be consenting adults undergoing various surgical procedures usually resulting in moderate-to-severe postoperative pain and treated with single-injection peripheral nerve blocks. Study inclusion will be proposed to eligible patients prior to surgery. If a patient desires study participation, written, informed consent will be obtained using a current UCSD IRB-approved ICF. The study population of interest includes women and men of all races, ethnicity, sexual identity, and socioeconomic status.

Preoperative Procedures. Following written, informed consent, the investigators will record baseline anthropometric information (age, sex, height, weight, current pain level). Participants will have their single-injection peripheral nerve block administered using ropivacaine 0.5% with epinephrine (standard at the enrolling institution) prior to undergoing their surgical procedure per standard of care. A "successful" regional block will be defined as sensory- and motor-block onset in all expected nerve distributions within the 30 minutes following the local anesthetic injection. Participants with a successful regional block and undergo the anticipated surgical procedure will be randomized and continue within the study.

Treatment Group Assignment. Each participant will be randomized to one of two treatment groups: Active (Experimental) or Sham treatment. There are sham devices produced that are identical to active devices, only they do not deliver electrical current. Randomization will be stratified by surgical procedure, in block sizes of 2. The computer-generated randomization list will be created by the University of California San Diego Investigational Drug Service in a 1:1 treatment group ratio assigned only after successful peripheral nerve block administration and the participant underwent the anticipated surgical procedure. The active and sham stimulators are indistinguishable in appearance, and therefore investigators, participants, and all clinical staff other than the individual who opens the randomization envelope and chooses a sham or active device will be masked to treatment group assignment for the duration of the data collection period.

Study intervention. The NSS-2 Bridge device will be affixed to the ear and activated prior to discharge from the recovery room (Experimental). There is currently no consensus regarding the placement on the ipsilateral or contralateral ear relative to the surgical procedure (if sided). Therefore, the investigators will apply the device to the side that the participant sleeps on least, to optimize comfort in bed and sleep.

Postoperative course. In addition to the experimental device and single-injection peripheral nerve block, participants will receive standard-of-care oral and intravenous postoperative analgesics which can include acetaminophen, ibuprofen, ketorolac, and opioids (this is surgeon- and patient-dependent). Therefore, all patients of this study-regardless of the treatment arm they are randomized to-will continue to receive current usual and customary analgesia: all will receive the same combination of acetaminophen, ibuprofen, ketorolac, opioids, and a single-injection peripheral nerve block as they would regardless of study participation. Prior to discharge, participants and their caretakers will be provided with verbal instructions regarding the care of the stimulator, and the telephone and pager numbers of an investigator available at all times during the first 5 days of treatment. The instructions for the stimulator are few: (1) participants can shower, but use a shower cap to cover the stimulator; (2) there are no controls so there is nothing that needs to be adjusted; (3) the device will run out of power after 5 days; (4) the investigators will call participants every day to answer any questions participants might have and describe how to remove the device as that time approaches.

Participants will be discharged when ready, as determined by standard criteria by the masked surgical service. Participants will be discharged home with their NSS-2 Bridge in situ and a prescription for immediate-release oral opioid, preferably oxycodone 5 mg tablets, taken for breakthrough pain. Participants will be contacted by telephone for end point collection beginning on postoperative day 1. The NSS-2 Bridge devices will be removed by patients or their caretakers at home on postoperative day 5. Similar to perineural catheters, this procedure encompasses simply removing the small dressings (the electrodes remain adhered to the dressings and therefore do not require a separate extraction step), removing the stimulator from behind the ear with simple traction, and discarding all components (these are disposable, single-use devices).

At the conclusion of the study, participants will be informed of the main results in lay-person language by either email or the U.S. Postal Service.

Study outcomes: This is an exploratory pilot study to assist in planning a subsequent definitive trial and the investigators therefore have no data analysis plan. The investigators will enroll convenience samples for each of the surgical procedures of up to 30 participants for each procedure and anticipate analyzing some surgical procedure separately from the others (hips, knees, breast, hernia/cholecystectomy, septoplasty). The two primary outcomes will be (1) the mean of the "average" pain recorded on postoperative days 1-5 measured with the Numeric Rating Scale ("average" pain is included in the Brief Pain Inventory pain domain); and (2) the cumulative opioids consumed from recovery room discharge until postoperative day 5, as measured in oral oxycodone equivalents.

ELIGIBILITY:
Inclusion Criteria:

1. undergoing one of these surgical procedures as a primary procedure (not revision):

   1. septoplasty [infraorbital nerve block]
   2. laparoscopic cholecystectomy [transversus abdominis nerve block]
   3. laparoscopic sleeve gastrectomy [transversus abdominis nerve block]
   4. non-mastectomy breast surgery [paravertebral nerve block]
   5. percutaneous nephrolithotomy [erector spinae plane nerve block]
   6. inguinal hernia repair [transversus abdominis nerve block]
   7. knee arthroplasty [adductor canal nerve block]
   8. hip arthroplasty [pericapsular nerve group block]
   9. shoulder acromioclavicular joint repair, labral repair, subacromial decompression, or Bankart repair (without rotator cuff repair) [interscalene nerve block]
   10. orthopedic hardware removal anticipated to be at least moderately painful postoperatively [various peripheral nerve blocks]
2. analgesic plan includes a single-injection peripheral nerve block with a long-acting local anesthetic [may be waived for hip arthroplasty]
3. age 18 years or older.

Exclusion Criteria:

1. concurrent use of another electric stimulator (e.g., cardiac pacemaker)
2. bleeding disorder
3. anticoagulation
4. skin abnormality at the treatment site
5. psoriasis vulgaris
6. morbid obesity as defined by a body mass index > 40
7. history of opioid abuse
8. inability to communicate with the investigators or hospital staff
9. pregnancy
10. bilateral or multi-stage surgical procedures
11. incarceration
12. chronic opioid or tramadol use (daily use within the 2 weeks prior to surgery and duration of use > 4 weeks)
13. neuro-muscular deficit of the surgical area/limb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2024-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD, Ms, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ilfeld BM, Abramson WB, Said ET, Sztain JF, Finneran JJ 4th, Griggs JL, Abdullah B, Jensen EJ, Schaar A, Wallace AM. Percutaneous auricular neuromodulation to treat pain after ambulatory breast surgery: A randomized, double-masked, sham-controlled pilot study. Can J Pain. 2025 Jul 10;9(1):2521117. doi: 10.1080/24740527.2025.2521117. eCollection 2025. PMID 40657450
- [Derived] Ilfeld BM, Finneran JJ 4th, Alexander B, Abramson WB, Sztain JF, Ball ST, Gonzales FB, Abdullah B, Cha BJ, Said ET. Percutaneous auricular neuromodulation (nerve stimulation) for the treatment of pain following total knee arthroplasty: a randomized, double-masked, sham-controlled pilot study. Reg Anesth Pain Med. 2025 Jan 7;50(1):26-35. doi: 10.1136/rapm-2023-105028. PMID 38388019
- [Derived] Ilfeld BM, Abramson WB, Alexander B, Sztain JF, Said ET, Broderick RC, Sandler BJ, Doucet JJ, Adams LM, Abdullah B, Cha BJ, Finneran JJ 4th. Percutaneous auricular neuromodulation (nerve stimulation) for the treatment of pain following cholecystectomy and hernia repair: a randomized, double-masked, sham-controlled pilot study. Reg Anesth Pain Med. 2024 Sep 2;49(9):628-634. doi: 10.1136/rapm-2024-105283. PMID 38388014

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Percutaneous Auricular Neuromodulation With NSS-2 Bridge | Sham Treatment
Started | 61 | 61
Completed | 60 | 60
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Percutaneous Auricular Neuromodulation With NSS-2 Bridge | Sham Treatment | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (15) | 62 (15) | 61 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 65
  Male | 28 | 27 | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120
Weight [Mean (Standard Deviation); unit: kg] | 79 (17) | 78 (16) | 78 (16)
Height [Mean (Standard Deviation); unit: cm] | 170 (11) | 170 (11) | 170 (11)
Body Mass Index [Mean (Standard Deviation); unit: kg / m^2] | 27 (5) | 27 (5) | 27 (5)

OUTCOME MEASURES:

1. Primary Outcome: AVERAGE Pain Measured With the Numeric Rating Scale First 5 Postoperative Days
Description: The numeric rating scale is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale. The outcome will the mean value of daily average pain scores measured with the Numeric Rating Scale. The primary outcome measure will be the mean value of the average daily pain measured on postoperative days 1-5.
Time Frame: The first 5 postoperative days
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Active Percutaneous Auricular Neuromodulation With NSS-2 Bridge | Sham Treatment
Number analyzed (Participants) | 60 | 60
units on a scale | 1 [0 to 3] | 3 [1 to 4]

2. Primary Outcome: Total OPIOID Consumption From Recovery Room Discharge Until the Data Collection Phone Call on Postoperative Day 5 (Measured in Oral Oxycodone Equivalents)
Description: Total opioid consumption from recovery room discharge until the data collection phone call on postoperative day 5 (measured in oral oxycodone equivalents).
Time Frame: Postoperative days 0-5
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Active Percutaneous Auricular Neuromodulation With NSS-2 Bridge | Sham Treatment
Number analyzed (Participants) | 60 | 60
mg | 5 [0 to 22.5] | 17.5 [0 to 60]

3. Secondary Outcome: AVERAGE Pain Measured With the Numeric Rating Scale
Description: The numeric rating scale is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale
Time Frame: Recorded on postoperative days 1-8 for the previous 24-hour period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Percutaneous Auricular Neuromodulation With NSS-2 Bridge | Sham Treatment
Number analyzed (Participants) | 60 | 60
units on a scale
  Day 1 | 2.3 (2) | 2.8 (2.3)
  Day 2 | 1.9 (2.2) | 3.3 (2.4)
  Day 3 | 1.8 (2.1) | 3 (2.5)
  Day 4 | 1.5 (1.8) | 2.7 (2)
  Day 5 | 1.5 (1.6) | 2.5 (1.9)
  Day 6 | 1.5 (1.6) | 2.3 (1.9)
  Day 7 | 1.5 (1.6) | 2.1 (1.9)
  Day 8 | 1.6 (1.9) | 1.8 (1.8)

4. Secondary Outcome: WORST (Highest or Maximum) Pain Measured With the Numeric Rating Scale
Description: as for outcome 3
Time Frame: Recorded on postoperative days 1-8 for the previous 24-hour period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Percutaneous Auricular Neuromodulation With NSS-2 Bridge | Sham Treatment
Number analyzed (Participants) | 60 | 60
units on a scale
  Day 1 | 4.3 (2.5) | 4.9 (2.8)
  Day 2 | 4 (3) | 5.5 (2.8)
  Day 3 | 3.7 (2.9) | 4.9 (2.6)
  Day 4 | 3 (2.5) | 4.4 (2.4)
  Day 5 | 3.1 (2.6) | 4.1 (2.6)
  Day 6 | 3.1 (2.7) | 4 (2.6)
  Day 7 | 3 (2.7) | 3.8 (2.8)
  Day 8 | 2.9 (3.1) | 3.2 (2.4)

5. Secondary Outcome: LEAST (Lowest or Minimum) Pain Measured With the Numeric Rating Scale
Description: as for outcome 3
Time Frame: Recorded on postoperative days 2, 4, 6, and 8 for the previous 24-hour period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Percutaneous Auricular Neuromodulation With NSS-2 Bridge | Sham Treatment
Number analyzed (Participants) | 60 | 60
units on a scale
  Day 2 | 1 (1.6) | 1.8 (1.9)
  Day 4 | .7 (1.3) | 1.2 (1.5)
  Day 6 | .6 (1.2) | 1.2 (1.5)
  Day 8 | .6 (1.2) | .9 (1.3)

6. Secondary Outcome: CURRENT Pain at the Time of the Data-collection Phone Call Measured With the Numeric Rating Scale
Description: as for outcome 3
Time Frame: Recorded on postoperative days 2, 4, 6, and 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Percutaneous Auricular Neuromodulation With NSS-2 Bridge | Sham Treatment
Number analyzed (Participants) | 60 | 60
units on a scale
  Day 2 | 1.5 (2) | 3 (2.6)
  Day 4 | 1.3 (1.8) | 2 (1.9)
  Day 6 | 1.3 (1.9) | 1.9 (2)
  Day 8 | 1.2 (1.8) | 1.6 (1.9)

7. Secondary Outcome: Opioid Consumption of the Previous 24 Hours (Measured in Oral Oxycodone Equivalents)
Description: Opioid consumption of the previous 24 hours (measured in oral oxycodone equivalents)
Time Frame: Recorded on postoperative days 1-8
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active Percutaneous Auricular Neuromodulation With NSS-2 Bridge | Sham Treatment
Number analyzed (Participants) | 60 | 60
mg
  Day 1 | 4.5 (8) | 8 (11.5)
  Day 2 | 6 (10) | 8 (12)
  Day 3 | 5 (10) | 8 (12)
  Day 4 | 4 (7.5) | 7.5 (12.5)
  Day 5 | 3 (5.5) | 7 (11.5)
  Day 6 | 2.5 (6) | 5 (9)
  Day 7 | 3 (6.5) | 4 (9)
  Day 8 | 3.5 (8) | 4 (8)

8. Secondary Outcome: Brief Pain Inventory, Short Form (Interference Subscale)
Description: The interference sub scale of the Brief Pain Inventory short form is an instrument specifically designed to assess pain's impact on physical and emotional functioning. It is comprised of 7 questions involving physical and emotional functioning using a 0-10 Likert scale [0=no interference, good;10=complete interference, bad]: general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life. The responses for these 7 questions are summed, resulting in a final scale of 0 (no interference=good) to 70 (complete interference=bad).
Time Frame: Recorded on postoperative days 2, 4, 6, and 8 for the previous 24-hour period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Percutaneous Auricular Neuromodulation With NSS-2 Bridge | Sham Treatment
Number analyzed (Participants) | 60 | 60
score on a scale
  Day 2 | 14 (17) | 23 (20)
  Day 4 | 11 (15) | 18 (17)
  Day 6 | 12 (17) | 17 (17)
  Day 8 | 9 (14) | 13 (16)

9. Secondary Outcome: Awakenings Due to Pain
Description: The number of times the participant awoke the previous night due to pain
Time Frame: Recorded on postoperative days 1-8 for the previous night
Measure: Median (Inter-Quartile Range); unit: number of awakenings
Arm/Group | Active Percutaneous Auricular Neuromodulation With NSS-2 Bridge | Sham Treatment
Number analyzed (Participants) | 60 | 60
number of awakenings
  Day 1 | 0 [0 to 0] | 0 [0 to 0]
  Day 2 | 0 [0 to 1] | 0 [0 to 1]
  Day 3 | 0 [0 to 0] | 0 [0 to .8]
  Day 4 | 0. [0 to 0.5] | 0 [0 to 1]
  Day 5 | 0 [0 to 0] | 0 [0 to 0.3]
  Day 6 | 0 [0 to 0] | 0 [0 to 1]
  Day 7 | 0 [0 to 0] | 0 [0 to 0]
  Day 8 | 0 [0 to 0] | 0 [0 to 1]

10. Secondary Outcome: Masking
Description: Patient queried if they thought they received active stimulation (entered as "1"), a sham device (entered as "0"), or are not sure (entered as "0.5")
Time Frame: Recorded on postoperative day 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Percutaneous Auricular Neuromodulation With NSS-2 Bridge | Sham Treatment
Number analyzed (Participants) | 60 | 60
score on a scale | .5 [.5 to 1] | .5 [.5 to 1]

11. Secondary Outcome: Hospitalization Duration Measured in Days
Description: Day relative to the day of surgery that patient was discharged from the hospital (e.g., same day is postoperative day 0, while the day following surgery is postoperative day 1)
Time Frame: Up to 2 weeks after surgery
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Active Percutaneous Auricular Neuromodulation With NSS-2 Bridge | Sham Treatment
Number analyzed (Participants) | 60 | 60
Days | .2 (.5) | .5 (.8)

12. Secondary Outcome: Tourniquet Duration
Description: Number of minutes the tourniquet was inflated
Time Frame: Intraoperative (within the operating room)
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Active Percutaneous Auricular Neuromodulation With NSS-2 Bridge | Sham Treatment
Number analyzed (Participants) | 60 | 60
Minutes | .8 (4.4) | 1.8 (9.5)

13. Secondary Outcome: Surgical Duration
Description: The time from surgical start to surgical stop measured in minutes and hours
Time Frame: Intraoperative (within the operating room)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Active Percutaneous Auricular Neuromodulation With NSS-2 Bridge | Sham Treatment
Number analyzed (Participants) | 60 | 60
minutes | 92.4 (41.5) | 89.3 (35.9)

ADVERSE EVENTS:
Time Frame: Within the 8 days following surgery
Arm/Group | Active Percutaneous Auricular Neuromodulation With NSS-2 Bridge | Sham Treatment
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT05521516/Prot_001.pdf